CLINICAL TRIAL: NCT03761225
Title: A Prospective, Multicenter, Randomized, Double Blind, Placebo-controlled, 2-parallel Groups, Phase 3 Study to Compare the Efficacy and Safety of Masitinib in Combination With Docetaxel to Placebo in Combination With Docetaxel in First Line Metastatic Castrate Resistant Prostate Cancer (mCRPC)
Brief Title: Masitinib Plus Docetaxel in Metastatic Castration-resistant Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AB12003
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Castrate Resistant Prostate Cancer
Keywords: metastatic castration-resistant prostate cancer; metastatic hormone-resistant prostate cancer; tyrosine kinase inhibitor; mCRPC; mHRPC
MeSH Terms: interventions — masitinib; Docetaxel; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Masitinib & docetaxel (Experimental): Participants receive masitinib (6 mg/kg/day), given orally twice daily, plus docetaxel 75 mg/m2 by intravenous infusion during 1 hour, once every 3 weeks (1 cycle = 21 days) for 6 cycles (8 to 10 cycles can be performed according to patient's tolerance) plus prednisone according to usual practice.
  Interventions: Drug: Masitinib; Drug: Docetaxel; Drug: Prednisone
- Placebo & docetaxel (Placebo Comparator): Participants receive placebo (6 mg/kg/day), given orally twice daily, plus docetaxel 75 mg/m2 by intravenous infusion during 1 hour, once every 3 weeks (1 cycle = 21 days) for 6 cycles (8 to 10 cycles can be performed according to patient's tolerance) plus prednisone according to usual practice.
  Interventions: Drug: Docetaxel; Drug: Prednisone; Drug: Placebo

INTERVENTIONS:
Drug: Masitinib
  Other Names: AB1010
  Arms: Masitinib & docetaxel
Drug: Docetaxel
Drug: Prednisone
Drug: Placebo
  Arms: Placebo & docetaxel

SUMMARY:
Study of masitinib plus docetaxel as first-line chemotherapy in men with metastatic castration-resistant prostate cancer.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the efficacy and safety of masitinib in combination with docetaxel and prednisone with respect to placebo in combination with docetaxel and prednisone in the treatment of first line metastatic Castrate Resistant Prostate Cancer (mCRPC). Approximately 580 patients will be randomized in 2 groups with a ratio 1:1. The primary outcome measure is progression free survival. Masitinib is a selective tyrosine kinase inhibitor that is thought to promote survival via modulation of immunostimulation-mediated anticancer effects and modulation of the tumor microenvironment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed metastatic Castrate Resistant Prostate Cancer (medical or surgical castration: androgens deprivation by GnHR agonist or antagonist or patient with surgical castration; hormonal castration confirmed biologically (testosterone < 0.5ng/ml) with one of the following criteria:

   * Pre-treated with abiraterone with documented progressive disease, OR
   * Indicated for initiating docetaxel treatment (e.g., widespread visceral disease or rapidly progressive disease).
2. Patient with evidence of progressive metastatic disease as assessed according to the Prostate Cancer Clinical Trials Working Group 2 (PCWG2) recommendations.
3. Patient with adequate organ function as per protocol

Exclusion Criteria:

1. Patient who has been previously treated with chemotherapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 714 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | From day of randomization to disease progression or death, assessed for a maximum of 60 months
  Progression Free Survival (PFS) is defined as the time from the randomization date until the date of earliest evidence of disease progression or death, for participants who progressed or died before subsequent cancer therapy. Disease progression will be assessed according to the Prostate Cancer Clinical Trials Working Group 2 (PCWG2) recommendations.

SECONDARY OUTCOMES:
Overall Survival | From day of randomization to death, assessed for a maximum of 60 months
  Overall survival (OS) is defined as time in months from the randomization date to the date of death due to any cause. If a patient is not known to have died, then OS will be censored at the date of last known date patient alive.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Spaeth, MD, Principal Investigator — Polyclinique d'oncologie de Gentilly, Nancy, France
Locations (9):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Canada
- Polyclinique d'oncologie de Gentilly, Nancy, France
- Sanjay Gandhi Post Graduate Institute of Medical Sciences, Lucknow, India
- Italy (3):
  - Centro di Riferimento Oncologico, Aviano
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- Universiti Malaya Medical Centre, Kuala Lumpur, Malaysia
- Russia (2):
  - Clinical Oncology Dispensary, Omsk
  - Clinic Andros LLC, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No